CLINICAL TRIAL: NCT02414620
Title: Efficacy of the Dental Vibe Unit for Use of Reduction or Elimination of Pain During Dental Anesthetic Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-40.7
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2012-07

CONDITIONS: Dental Pain
Keywords: Efficacy; Dental Vibe Unit; Reduction; Elimination; Dental Anesthetic Injection
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dental Vibe (Experimental): New oscillating device for reduction in pain during dental anesthesia
  Interventions: Device: Generation II Dental Vibe Unit

INTERVENTIONS:
Device: Generation II Dental Vibe Unit — . The Dental Vibe emits strong pulsed vibration which is transmitted via a silicone mouth piece to mucosal tissue.

SUMMARY:
The purpose of the research was to test the efficacy of the Dental Vibe Injection Comfort System. The study was conducted by faculty to have students as subjects to see if there are any differences in the comfort level of an ASA injection given on one side with topical anesthesia and lidocaine 1:100,000 with epinephrine using a standard syringe, and the other side uing the Dental Vibe, topical anesthesia and lidocaine 1:100,000 with epinephrine and a standard syringe. The Dental Vibe emits strong pulsed vibration which is transmitted via a silicone mouth piece to mucosal tissue. This in turn interferes with, blocks or reduces the perception of pain from the injection for the patient. It is stated that this phenomenon is achieved due to the "gate theory" of neuronal activity. There are also likely, distraction and placebo effects that contribute to the devices' efficacy.

DETAILED DESCRIPTION:
Subjects were in groups of 3-4 for 2 ½ hours where 1 subject will be the operator delivering injection, 1 subject will be the assistant, and 1 subject was the patient receiving the injection. It was all be conducted in the pre-clinical local anesthesia rotation in a clinical setting. OSHA regulations will be followed and supplies was provided for subjects.

Using standard syringe, the operator assembled a 27 gauge short needle and load a 2% lidocaine 1:100,000 epi cartridge. Gauze was applied to the area of the upper right muccobuccal fold, where the penetration site of the ASA injection was administered. Small amount of topical will be placed at penetration site and left for approximately one minute. The subject posing as the operator obtained a retraction method using a mouth mirror. The ASA injection technique was then be applied and 1/3 cartridge of solution will be administered at the deposition site.

Immediately after, using same standard syringe and remaining anesthestic cartridge, the operator replaced the 27 gauge short needle. Gauze was applied to the area of the upper left muccobuccal fold, where the penetration site of the ASA injection was administered. Small amount of topical was placed at penetration site and left for approximately one minute. The subject posing as the operator will obtain a retraction method using the Dental Vibe Unit, turn the device on and kept active for 3-5 seconds prior to, during, and after needle penetration. The ASA injection technique was applied and 1/3 cartridge of solution was administered at the deposition site.

The ASA injection technique had a penetration site into the muccobuccal fold above or in between the maxillary canine and maxillary first pre-molar. The depth of penetration was initially 3 mm into soft tissue, and then the needle was slowly advanced an additional 2 mm or until bone was gently reached. Anesthesia was then deposited at a rate of ¼ cartridge / 15 seconds. An aspiration test was given, which then confirmed that anesthesia was not being deposited into a blood vessel. Once 1/3 cartridge was dispensed, needle was then removed from site.

An evaluation then was given to the subject posing as the patient. The subjects was carefully observed for appropriate site preparation, injection technique, proper placement of mouth mirror, and proper placement of Dental Vibe Unit.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be first and second year students giving their injections during their anesthesia rotation. Subjects are not being actively recruited.

Exclusion Criteria:

* Students will be given the option to voluntarily participate in this study during their normally scheduled anesthesia rotation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
reduction of pain in dental anesthesia | 15 min